CLINICAL TRIAL: NCT05619601
Title: Gender Differences in Prevention Strategies and Therapeutic Adherence After Acute Myocardial Infarction - GENAMI PREVENTION
Brief Title: Gender Differences in Prevention Strategies and Therapeutic Adherence After Acute Myocardial Infarction
Acronym: GENAMI
Status: Active, not recruiting | Type: Observational
Sponsor: Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Héctor Bueno, Principal Investigator, Spanish Society of Cardiology
Other Study IDs: 0099-2022-OBS
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Gender Differences; Adherence, Medication; Therapeutic Adherence; Type 1 Acute Myocardial Infarction
Keywords: Gender; Adherence; Acute myocardial infarction
MeSH Terms: conditions — Medication Adherence; Treatment Adherence and Compliance; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 500 women: 500 women discharged alive after a hospitalization for a type 1 acute myocardial infarction with significant coronary artery disease.
- 500 men: 500 age (±2 years) and ECG (STEMI/NSTEMI) locally matched men discharged alive after a hospitalization for a type 1 acute myocardial infarction with significant coronary artery disease.

SUMMARY:
PARTICIPANT CENTERS: 25 hospitals managing routinely acute myocardial infarction (AMI) and representing different regions from Spain will be invited to participate.

GENERAL OBJECTIVE: To evaluate if there are differences in the level of adherence to recommended secondary prevention therapies (pharmacological and non-pharmacological) between women and men surviving a type 1 acute myocardial infarction (with obstructive coronary artery disease), its potential consequences, and the potential factors related to that difference, if present.

DESIGN:

Prospective, matched cohort study of patients hospitalized for a type 1 acute myocardial infarction with evidence of obstructive coronary artery disease who are discharged home alive. Women will be enrolled first, ideally in a consecutive manner, as they are the focus of the study. Men will be recruited subsequently as the comparison group, with 1:1 matching for age and ECG presentation. Matching will be performed locally, in each study site (hospital). All patients will undergo 1-year follow-up with clinical and therapeutic adherence evaluation.

- Reference cohort: 500 women discharged alive after a hospitalization for a type 1 acute myocardial infarction with significant coronary artery disease.

- Comparator cohort: 500 age (±2 years) and ECG (ST-segment elevation acute myocardial infarction (STEMI) / non-ST-segment elevation acute myocardial infarction (NSTEMI)) locally matched men discharged alive after a hospitalization for a type 1 acute myocardial infarction with significant coronary artery disease.

DETAILED DESCRIPTION:
OBJECTIVES

General objective: To evaluate if there are differences in the level of adherence to recommended secondary prevention therapies (pharmacological and non-pharmacological) between women and men surviving a type 1 acute myocardial infarction (with obstructive coronary artery disease), its potential consequences, and the potential factors related to that difference, if present.

Specific objectives: To compare between women and men:

1) The adherence to recommended secondary prevention therapies at 6 months and 12 months measured as the:

1a. Proportion of patients adherent to all recommended pharmacological secondary prevention therapies at 6 and 12 months.

1b. Proportion of patients adherent to all recommended non-pharmacological secondary prevention therapies at 6 and 12 months.

2) The relationship of the adherence with control of risk factors, clinical outcomes, and use of healthcare resources.

2a. The proportion of patients with optimal control of all cardiovascular risk factors at 6 and 12 months.

2b. The incidence of clinical outcomes at 6 and 12 months. 2c. The cumulative use of healthcare resources and cost after discharge.

3) To assess the factors associated with non-adherence to recommended secondary prevention therapies, with special emphasis to socioeconomic factors and gender issues.

STUDY DESIGN

DESIGN:

Prospective, matched cohort study of patients hospitalized for a type 1 acute myocardial infarction with evidence of obstructive coronary artery disease who are discharged home alive. Women will be enrolled first, ideally in a consecutive manner, as they are the focus of the study. Men will be recruited subsequently as the comparison group, with 1:1 matching for age and ECG presentation. Matching will be performed locally, in each study site (hospital). All patients will undergo 1-year follow-up with clinical and therapeutic adherence evaluation.

RECRUITMENT:

Participant centers:

25 hospitals managing routinely acute myocardial infarction and representing different regions from Spain will be invited to participate.

Patient recruitment:

All consecutive women fulfilling all inclusion criteria and without exclusion criteria surviving the index hospitalization will be invited to participate. Subsequently, men with inclusion criteria and without exclusion criteria, matched for age and ECG presentation, will be recruited.

STATISTICAL ANALYSIS:

A minimum sample size of 820 participants (410 per group) was estimated for an expected relative difference in recommendations compliance of the all-or-none composite primary outcome of 20%. An α error of 0.05 and a β error of 0.20 were considered for the sample size. The recommendations compliance was estimated as 42% for women and 52% for men. With the consideration of 20% of lost to follow-up (discontinuations) the total sample size is 984 patients, which is rounded out to 1000 patients (500 women and 500 men). To increase regional representation and allow exploration of potential regional variability, 25 hospitals from all regions in Spain (17 Autonomous Communities) will be invited to participate.

For the description of continuous variables, mean and standard deviation, or median and interquartile range will be used for Gaussian and non-normal distributions, respectively. For describing categorical variables, frequencies and percentages per category will be used. Categorical variables will be compared using the chi2 test, whilst continuous variables will be compared using the student t test.

Logistic regression models will be used to evaluate differences in binary outcomes between women and men (in hospital acute myocardial infarction management, post discharge myocardial infarction management). All subjects will be assumed to have a fixed follow-up (12±1 month). Multivariate adjusted models will be used to address any potential confounding in the associations between sex and each of the outcomes. Covariates will be selected based on their pre-defined clinical value and the unbalances observed across groups in the univariate analyses. Linear, multinomial or ordinal regression models would be used in case of continuous, categorical, or ordinal outcomes, respectively.

In addition to the models evaluating the association between sex and outcomes, a predictive model will be conducted to set predictors for the following outcomes:

1. a composite of all preventive therapies (all-or-nothing for diet, physical activity, P2Y12 inhibitors, statins, and beta blockers or angiotensin converting enzyme inhibitors [if prescribed at discharge]), and
2. each group of preventive interventions (drugs, cardiac rehab, diet, physical activity) Candidate predictors are classified as biological factors (age, sex, risk factors, comorbidities), disease-related (type of myocardial infarction: ST-segment elevation acute myocardial infarction (STEMI) / non-ST-segment elevation acute myocardial infarction (NSTEMI), left ventricular ejection fraction, number of vessels…), pharmacological factors (daily number of drugs, daily number of doses, specific drugs), socio-economic factors (zip code, education level, employment status, wages…) and specific gender issues (family responsibilities, work conciliation…). Special consideration will be given to age due to the high figures of in-hospital mortality in young women.

For women-specific analysis, female specific factors (menarche age, pregnancies, gestational diabetes, menopause…) will be considered.

It will be used the Clinical Outcomes, HEalthcare REsource UtilizatioN, and relaTed costs (COHERENT) model to study the hospital-related healthcare resources (emergency department visits, specialist visits, re-hospitalizations and urgent procedures) and costs.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for a type 1 acute myocardial infarction (detection of a rise and/or fall of troponin c value above the 99th percentile upper reference limit (URL) and with at least one of the followings: symptoms of acute myocardial ischemia; new ischaemic ECG changes; development of pathological Q waves; imaging evidence of new loss of viable myocardium or new regional wall motion abnormality in a patterns consistent with an ischaemic aetiology; identification of a coronary thrombus by angiography including intracoronary imaging)
* Presence of obstructive coronary artery disease (CAD) (i.e. coronary artery stenosis ≥50%)
* Age >18 years. No maximal age limit applies
* Signed informed consent

Exclusion Criteria:

* Terminal disease (expected survival <12 months)
* Unavailable for 12-month follow-up (i.e.: living abroad, social situation…)
* Does not speak Spanish
* Major active comorbidity (severe renal or liver failure, active cancer requiring chemotherapy…), interfering with regular post-myocardial infarction management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective, matched cohort study of patients hospitalized for a type 1 AMI with evidence of obstructive coronary artery disease who are discharged home alive. Women will be enrolled first, ideally in a consecutive manner, as they are the focus of the study. Men will be recruited subsequently as the comparison group, with 1:1 matching for age and ECG presentation. Matching will be performed locally, in each study site (hospital). All patients will undergo 1-year follow-up with clinical and therapeutic adherence evaluation.
  Reference cohort: 500 women discharged alive after a hospitalization for a type 1 AMI with significant CAD.
  Comparator cohort: 500 age (±2 years) and ECG (STEMI/NSTEMI) locally matched men discharged alive after a hospitalization for a type 1 AMI with significant CAD.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of adherence to all secondary cardiovascular prevention recommendations at 12 months after discharge | 12 months
  The composite is built as an all-or-nothing response to an adherence ≥80% in all prescribed components of the endpoint: pharmacological therapies (MMAS-8), diet, physical activity and participation in a cardiac rehabilitation program. Adherence will be defined as having at least 80% compliance with all cardiovascular prevention recommendations; drugs, cardiac rehabilitation program, diet and physical activity)
Pharmacological primary endpoint | 12 months
  Outcome of adherence to pharmacological therapies (MMAS-8) 12 months after discharge
Non-pharmacological primary endpoint | 12 months
  Composite outcome of adherence to non-pharmacological secondary cardiovascular prevention recommendations 12 months after discharge, including diet, physical activity and participation in cardiac rehabilitation programs

SECONDARY OUTCOMES:
Pharmacological primary endpoint | 6 months
  Outcome of adherence to pharmacological therapies (MMAS-8) 6 months after discharge
Non-pharmacological primary endpoint | 6 months
  Composite outcome of adherence to non-pharmacological secondary cardiovascular prevention recommendations 6 months after discharge, including diet, physical activity and participation in cardiac rehabilitation programs

CONTACTS AND LOCATIONS:
Overall Officials: Hector Bueno, MD, PhD, Principal Investigator — Hospital Universitario 12 de Octubre, Madrid
Locations (25):
- Spain (25):
  - Hospital Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Universitari Son Espases, Palma de Mallorca, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Álvaro Cunqueiro de Vigo, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Complejo Hospitalario Universitario de Canarias, La Laguna, San Cristóbal de La Laguna, Tenerife
  - Hospital Universitario de Áraba/Txagorritxu, Vitoria-Gasteiz, Vitoria
  - Hospital Universitario de Basurto, Bilbao, Vizcaya
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario Vall´d Hebron, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Complejo Asistencial Universitario de León, León
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Complejo Hospitalario de Toledo, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nowbar AN, Gitto M, Howard JP, Francis DP, Al-Lamee R. Mortality From Ischemic Heart Disease. Circ Cardiovasc Qual Outcomes. 2019 Jun;12(6):e005375. doi: 10.1161/CIRCOUTCOMES.118.005375. Epub 2019 Jun 4. PMID 31163980
- [Background] Maas AHEM, Rosano G, Cifkova R, Chieffo A, van Dijken D, Hamoda H, Kunadian V, Laan E, Lambrinoudaki I, Maclaran K, Panay N, Stevenson JC, van Trotsenburg M, Collins P. Cardiovascular health after menopause transition, pregnancy disorders, and other gynaecologic conditions: a consensus document from European cardiologists, gynaecologists, and endocrinologists. Eur Heart J. 2021 Mar 7;42(10):967-984. doi: 10.1093/eurheartj/ehaa1044. PMID 33495787
- [Background] Jagannathan R, Patel SA, Ali MK, Narayan KMV. Global Updates on Cardiovascular Disease Mortality Trends and Attribution of Traditional Risk Factors. Curr Diab Rep. 2019 Jun 20;19(7):44. doi: 10.1007/s11892-019-1161-2. PMID 31222515
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] Yeh RW, Sidney S, Chandra M, Sorel M, Selby JV, Go AS. Population trends in the incidence and outcomes of acute myocardial infarction. N Engl J Med. 2010 Jun 10;362(23):2155-65. doi: 10.1056/NEJMoa0908610. PMID 20558366
- [Background] Neumann JT, Gossling A, Sorensen NA, Blankenberg S, Magnussen C, Westermann D. Temporal trends in incidence and outcome of acute coronary syndrome. Clin Res Cardiol. 2020 Sep;109(9):1186-1192. doi: 10.1007/s00392-020-01612-1. Epub 2020 Feb 7. PMID 32034482
- [Background] Chi GC, Kanter MH, Li BH, Qian L, Reading SR, Harrison TN, Jacobsen SJ, Scott RD, Cavendish JJ, Lawrence JM, Tartof SY, Reynolds K. Trends in Acute Myocardial Infarction by Race and Ethnicity. J Am Heart Assoc. 2020 Mar 3;9(5):e013542. doi: 10.1161/JAHA.119.013542. Epub 2020 Mar 2. PMID 32114888
- [Background] Goldberg RJ, Tisminetzky M, Tran HV, Yarzebski J, Lessard D, Gore JM. Decade Long Trends (2001-2011) in the Incidence Rates of Initial Acute Myocardial Infarction. Am J Cardiol. 2019 Jan 15;123(2):206-211. doi: 10.1016/j.amjcard.2018.10.002. Epub 2018 Oct 19. PMID 30409411
- [Background] Bangalore S, Fonarow GC, Peterson ED, Hellkamp AS, Hernandez AF, Laskey W, Peacock WF, Cannon CP, Schwamm LH, Bhatt DL; Get with the Guidelines Steering Committee and Investigators. Age and gender differences in quality of care and outcomes for patients with ST-segment elevation myocardial infarction. Am J Med. 2012 Oct;125(10):1000-9. doi: 10.1016/j.amjmed.2011.11.016. Epub 2012 Jun 27. PMID 22748404
- [Background] Bossard M, Latifi Y, Fabbri M, Kurmann R, Brinkert M, Wolfrum M, Berte B, Cuculi F, Toggweiler S, Kobza R, Chamberlain AM, Moccetti F. Increasing Mortality From Premature Coronary Artery Disease in Women in the Rural United States. J Am Heart Assoc. 2020 May 5;9(9):e015334. doi: 10.1161/JAHA.119.015334. Epub 2020 Apr 22. PMID 32316803
- [Background] Arora S, Stouffer GA, Kucharska-Newton AM, Qamar A, Vaduganathan M, Pandey A, Porterfield D, Blankstein R, Rosamond WD, Bhatt DL, Caughey MC. Twenty Year Trends and Sex Differences in Young Adults Hospitalized With Acute Myocardial Infarction. Circulation. 2019 Feb 19;139(8):1047-1056. doi: 10.1161/CIRCULATIONAHA.118.037137. PMID 30586725
- [Background] Wu WY, Berman AN, Biery DW, Blankstein R. Recent trends in acute myocardial infarction among the young. Curr Opin Cardiol. 2020 Sep;35(5):524-530. doi: 10.1097/HCO.0000000000000781. PMID 32694263
- [Background] Rodriguez-Padial L, Fernandez-Perez C, Bernal JL, Anguita M, Sambola A, Fernandez-Ortiz A, Elola FJ. Differences in in-hospital mortality after STEMI versus NSTEMI by sex. Eleven-year trend in the Spanish National Health Service. Rev Esp Cardiol (Engl Ed). 2021 Jun;74(6):510-517. doi: 10.1016/j.rec.2020.04.017. Epub 2020 Jun 16. English, Spanish. PMID 32561143
- [Background] Cortes-Beringola A, Fitzsimons D, Pelliccia A, Moreno G, Martin-Asenjo R, Bueno H. Planning secondary prevention: Room for improvement. Eur J Prev Cardiol. 2017 Jun;24(3_suppl):22-28. doi: 10.1177/2047487317704954. PMID 28618903
- [Background] Mehta LS, Beckie TM, DeVon HA, Grines CL, Krumholz HM, Johnson MN, Lindley KJ, Vaccarino V, Wang TY, Watson KE, Wenger NK; American Heart Association Cardiovascular Disease in Women and Special Populations Committee of the Council on Clinical Cardiology, Council on Epidemiology and Prevention, Council on Cardiovascular and Stroke Nursing, and Council on Quality of Care and Outcomes Research. Acute Myocardial Infarction in Women: A Scientific Statement From the American Heart Association. Circulation. 2016 Mar 1;133(9):916-47. doi: 10.1161/CIR.0000000000000351. Epub 2016 Jan 25. PMID 26811316
- [Background] Woodward M. Cardiovascular Disease and the Female Disadvantage. Int J Environ Res Public Health. 2019 Apr 1;16(7):1165. doi: 10.3390/ijerph16071165. PMID 30939754
- [Background] Hyun KK, Redfern J, Patel A, Peiris D, Brieger D, Sullivan D, Harris M, Usherwood T, MacMahon S, Lyford M, Woodward M. Gender inequalities in cardiovascular risk factor assessment and management in primary healthcare. Heart. 2017 Apr;103(7):492-498. doi: 10.1136/heartjnl-2016-310216. Epub 2017 Mar 1. PMID 28249996
- [Background] Young L, Cho L. Unique cardiovascular risk factors in women. Heart. 2019 Nov;105(21):1656-1660. doi: 10.1136/heartjnl-2018-314268. Epub 2019 Jul 17. PMID 31315936
- [Background] Gao Z, Chen Z, Sun A, Deng X. Gender differences in cardiovascular disease. Medicine in Novel Technology and Devices. 2019;4:100025.
- [Background] EUGenMed Cardiovascular Clinical Study Group; Regitz-Zagrosek V, Oertelt-Prigione S, Prescott E, Franconi F, Gerdts E, Foryst-Ludwig A, Maas AH, Kautzky-Willer A, Knappe-Wegner D, Kintscher U, Ladwig KH, Schenck-Gustafsson K, Stangl V. Gender in cardiovascular diseases: impact on clinical manifestations, management, and outcomes. Eur Heart J. 2016 Jan 1;37(1):24-34. doi: 10.1093/eurheartj/ehv598. Epub 2015 Nov 3. No abstract available. PMID 26530104
- [Background] Regitz-Zagrosek V, Kararigas G. Mechanistic Pathways of Sex Differences in Cardiovascular Disease. Physiol Rev. 2017 Jan;97(1):1-37. doi: 10.1152/physrev.00021.2015. PMID 27807199
- [Background] Gerdts E, Regitz-Zagrosek V. Sex differences in cardiometabolic disorders. Nat Med. 2019 Nov;25(11):1657-1666. doi: 10.1038/s41591-019-0643-8. Epub 2019 Nov 7. PMID 31700185
- [Background] Peters SA, Woodward M. Women's reproductive factors and incident cardiovascular disease in the UK Biobank. Heart. 2018 Jul;104(13):1069-1075. doi: 10.1136/heartjnl-2017-312289. Epub 2018 Jan 15. PMID 29335253
- [Background] Agarwala A, Michos ED, Samad Z, Ballantyne CM, Virani SS. The Use of Sex-Specific Factors in the Assessment of Women's Cardiovascular Risk. Circulation. 2020 Feb 18;141(7):592-599. doi: 10.1161/CIRCULATIONAHA.119.043429. Epub 2020 Feb 17. PMID 32065772
- [Background] Torris C, Bjornnes AK. Duration of Lactation and Maternal Risk of Metabolic Syndrome: A Systematic Review and Meta-Analysis. Nutrients. 2020 Sep 5;12(9):2718. doi: 10.3390/nu12092718. PMID 32899507
- [Background] Hayward CS, Kelly RP, Collins P. The roles of gender, the menopause and hormone replacement on cardiovascular function. Cardiovasc Res. 2000 Apr;46(1):28-49. doi: 10.1016/s0008-6363(00)00005-5. No abstract available. PMID 10727651
- [Background] Parker WH, Jacoby V, Shoupe D, Rocca W. Effect of bilateral oophorectomy on women's long-term health. Womens Health (Lond). 2009 Sep;5(5):565-76. doi: 10.2217/whe.09.42. PMID 19702455
- [Background] Smith SB, Geske JB, Kathuria P, Cuttica M, Schimmel DR, Courtney DM, Waterer GW, Wunderink RG. Analysis of National Trends in Admissions for Pulmonary Embolism. Chest. 2016 Jul;150(1):35-45. doi: 10.1016/j.chest.2016.02.638. Epub 2016 Feb 18. PMID 26905364
- [Background] Rosvall M, Gerward S, Engstrom G, Hedblad B. Income and short-term case fatality after myocardial infarction in the whole middle-aged population of Malmo, Sweden. Eur J Public Health. 2008 Oct;18(5):533-8. doi: 10.1093/eurpub/ckn059. Epub 2008 Jul 11. PMID 18621776
- [Background] Coughlin SS, Young L. Social Determinants of Myocardial Infarction Risk and Survival: A Systematic Review. Eur j Cardiovasc Res. 2020;1(1):10.31487/j.ejcr.2020.01.02. doi: 10.31487/j.ejcr.2020.01.02. Epub 2020 Sep 18. PMID 33089252
- [Background] Deguen S, Lalloue B, Bard D, Havard S, Arveiler D, Zmirou-Navier D. A small-area ecologic study of myocardial infarction, neighborhood deprivation, and sex: a Bayesian modeling approach. Epidemiology. 2010 Jul;21(4):459-66. doi: 10.1097/EDE.0b013e3181e09925. PMID 20489648
- [Background] Koopman C, van Oeffelen AA, Bots ML, Engelfriet PM, Verschuren WM, van Rossem L, van Dis I, Capewell S, Vaartjes I. Neighbourhood socioeconomic inequalities in incidence of acute myocardial infarction: a cohort study quantifying age- and gender-specific differences in relative and absolute terms. BMC Public Health. 2012 Aug 7;12:617. doi: 10.1186/1471-2458-12-617. PMID 22870916
- [Background] Peterson PN. JAHA Spotlight on Psychosocial Factors and Cardiovascular Disease. J Am Heart Assoc. 2020 May 5;9(9):e017112. doi: 10.1161/JAHA.120.017112. Epub 2020 Apr 28. No abstract available. PMID 32342721
- [Background] Greaney JL, Koffer RE, Saunders EFH, Almeida DM, Alexander LM. Self-Reported Everyday Psychosocial Stressors Are Associated With Greater Impairments in Endothelial Function in Young Adults With Major Depressive Disorder. J Am Heart Assoc. 2019 Feb 19;8(4):e010825. doi: 10.1161/JAHA.118.010825. PMID 30741602
- [Background] Rozanski A, Blumenthal JA, Kaplan J. Impact of psychological factors on the pathogenesis of cardiovascular disease and implications for therapy. Circulation. 1999 Apr 27;99(16):2192-217. doi: 10.1161/01.cir.99.16.2192. PMID 10217662
- [Background] Greaney JL, Surachman A, Saunders EFH, Alexander LM, Almeida DM. Greater Daily Psychosocial Stress Exposure is Associated With Increased Norepinephrine-Induced Vasoconstriction in Young Adults. J Am Heart Assoc. 2020 May 5;9(9):e015697. doi: 10.1161/JAHA.119.015697. Epub 2020 Apr 28. PMID 32340506
- [Background] Mittleman MA, Maclure M, Sherwood JB, Mulry RP, Tofler GH, Jacobs SC, Friedman R, Benson H, Muller JE. Triggering of acute myocardial infarction onset by episodes of anger. Determinants of Myocardial Infarction Onset Study Investigators. Circulation. 1995 Oct 1;92(7):1720-5. doi: 10.1161/01.cir.92.7.1720. PMID 7671353
- [Background] Nabi H, Kivimaki M, Batty GD, Shipley MJ, Britton A, Brunner EJ, Vahtera J, Lemogne C, Elbaz A, Singh-Manoux A. Increased risk of coronary heart disease among individuals reporting adverse impact of stress on their health: the Whitehall II prospective cohort study. Eur Heart J. 2013 Sep;34(34):2697-705. doi: 10.1093/eurheartj/eht216. Epub 2013 Jun 26. PMID 23804585
- [Background] Molarius A, Metsini A. Domestic Work, Self-Reported Diagnosed Depression and Related Costs among Women and Men-Results from a Population-Based Study in Sweden. Int J Environ Res Public Health. 2021 Sep 16;18(18):9778. doi: 10.3390/ijerph18189778. PMID 34574699
- [Background] Lundberg U, Mardberg B, Frankenhaeuser M. The total workload of male and female white collar workers as related to age, occupational level, and number of children. Scand J Psychol. 1994 Dec;35(4):315-27. doi: 10.1111/j.1467-9450.1994.tb00956.x. PMID 7809584
- [Background] Vaccarino V, Shah AJ, Rooks C, Ibeanu I, Nye JA, Pimple P, Salerno A, D'Marco L, Karohl C, Bremner JD, Raggi P. Sex differences in mental stress-induced myocardial ischemia in young survivors of an acute myocardial infarction. Psychosom Med. 2014 Apr;76(3):171-80. doi: 10.1097/PSY.0000000000000045. PMID 24608039
- [Background] Rossello X, Mas-Llado C, Pocock S, Vicent L, van de Werf F, Chin CT, Danchin N, Lee SWL, Medina J, Huo Y, Bueno H. Sex differences in mortality after an acute coronary syndrome increase with lower country wealth and higher income inequality. Rev Esp Cardiol (Engl Ed). 2022 May;75(5):392-400. doi: 10.1016/j.rec.2021.05.006. Epub 2021 Jun 24. English, Spanish. PMID 34175245
- [Background] Lichtman JH, Froelicher ES, Blumenthal JA, Carney RM, Doering LV, Frasure-Smith N, Freedland KE, Jaffe AS, Leifheit-Limson EC, Sheps DS, Vaccarino V, Wulsin L; American Heart Association Statistics Committee of the Council on Epidemiology and Prevention and the Council on Cardiovascular and Stroke Nursing. Depression as a risk factor for poor prognosis among patients with acute coronary syndrome: systematic review and recommendations: a scientific statement from the American Heart Association. Circulation. 2014 Mar 25;129(12):1350-69. doi: 10.1161/CIR.0000000000000019. Epub 2014 Feb 24. PMID 24566200
- [Background] Smolderen KG, Strait KM, Dreyer RP, D'Onofrio G, Zhou S, Lichtman JH, Geda M, Bueno H, Beltrame J, Safdar B, Krumholz HM, Spertus JA. Depressive symptoms in younger women and men with acute myocardial infarction: insights from the VIRGO study. J Am Heart Assoc. 2015 Apr 2;4(4):e001424. doi: 10.1161/JAHA.114.001424. PMID 25836055
- [Background] Rossi AM, Pilote L. Let's Talk About Sex...and Gender! Circ Cardiovasc Qual Outcomes. 2016 Feb;9(2 Suppl 1):S100-1. doi: 10.1161/CIRCOUTCOMES.116.002660. No abstract available. PMID 26908854
- [Background] Wu J, Gale CP, Hall M, Dondo TB, Metcalfe E, Oliver G, Batin PD, Hemingway H, Timmis A, West RM. Editor's Choice - Impact of initial hospital diagnosis on mortality for acute myocardial infarction: A national cohort study. Eur Heart J Acute Cardiovasc Care. 2018 Mar;7(2):139-148. doi: 10.1177/2048872616661693. Epub 2016 Aug 29. PMID 27574333
- [Background] Bugiardini R, Ricci B, Cenko E, Vasiljevic Z, Kedev S, Davidovic G, Zdravkovic M, Milicic D, Dilic M, Manfrini O, Koller A, Badimon L. Delayed Care and Mortality Among Women and Men With Myocardial Infarction. J Am Heart Assoc. 2017 Aug 21;6(8):e005968. doi: 10.1161/JAHA.117.005968. PMID 28862963
- [Background] Ahmed B, Dauerman HL. Women, bleeding, and coronary intervention. Circulation. 2013 Feb 5;127(5):641-9. doi: 10.1161/CIRCULATIONAHA.112.108290. No abstract available. PMID 23381962
- [Background] Damluji AA, van Diepen S, Katz JN, Menon V, Tamis-Holland JE, Bakitas M, Cohen MG, Balsam LB, Chikwe J; American Heart Association Council on Clinical Cardiology; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Cardiovascular Surgery and Anesthesia; and Council on Cardiovascular and Stroke Nursing. Mechanical Complications of Acute Myocardial Infarction: A Scientific Statement From the American Heart Association. Circulation. 2021 Jul 13;144(2):e16-e35. doi: 10.1161/CIR.0000000000000985. Epub 2021 Jun 15. PMID 34126755
- [Background] Kuehnemund L, Koeppe J, Feld J, Wiederhold A, Illner J, Makowski L, Gerss J, Reinecke H, Freisinger E. Gender differences in acute myocardial infarction-A nationwide German real-life analysis from 2014 to 2017. Clin Cardiol. 2021 Jul;44(7):890-898. doi: 10.1002/clc.23662. Epub 2021 Jun 1. PMID 34075604
- [Background] Matetic A, Shamkhani W, Rashid M, Volgman AS, Van Spall HGC, Coutinho T, Mehta LS, Sharma G, Parwani P, Mohamed MO, Mamas MA. Trends of Sex Differences in Clinical Outcomes After Myocardial Infarction in the United States. CJC Open. 2021 Jul 1;3(12 Suppl):S19-S27. doi: 10.1016/j.cjco.2021.06.012. eCollection 2021 Dec. PMID 34993430
- [Background] Eindhoven DC, Hilt AD, Zwaan TC, Schalij MJ, Borleffs CJW. Age and gender differences in medical adherence after myocardial infarction: Women do not receive optimal treatment - The Netherlands claims database. Eur J Prev Cardiol. 2018 Jan;25(2):181-189. doi: 10.1177/2047487317744363. Epub 2017 Nov 22. PMID 29164916
- [Background] Hyun K, Negrone A, Redfern J, Atkins E, Chow C, Kilian J, Rajaratnam R, Brieger D. Gender Difference in Secondary Prevention of Cardiovascular Disease and Outcomes Following the Survival of Acute Coronary Syndrome. Heart Lung Circ. 2021 Jan;30(1):121-127. doi: 10.1016/j.hlc.2020.06.026. Epub 2020 Sep 2. PMID 32888821
- [Background] Gulati M, Hendry C, Parapid B, Mulvagh SL. Why We Need Specialised Centres for Women's Hearts: Changing the Face of Cardiovascular Care for Women. Eur Cardiol. 2021 Dec 9;16:e52. doi: 10.15420/ecr.2021.49. eCollection 2021 Feb. PMID 35024054
- [Background] Smolina K, Ball L, Humphries KH, Khan N, Morgan SG. Sex Disparities in Post-Acute Myocardial Infarction Pharmacologic Treatment Initiation and Adherence: Problem for Young Women. Circ Cardiovasc Qual Outcomes. 2015 Nov;8(6):586-92. doi: 10.1161/CIRCOUTCOMES.115.001987. Epub 2015 Oct 13. PMID 26462876
- [Background] Hao Y, Liu J, Liu J, Yang N, Smith SC Jr, Huo Y, Fonarow GC, Ge J, Taubert KA, Morgan L, Zhou M, Xing Y, Ma CS, Han Y, Zhao D. Sex Differences in In-Hospital Management and Outcomes of Patients With Acute Coronary Syndrome. Circulation. 2019 Apr 9;139(15):1776-1785. doi: 10.1161/CIRCULATIONAHA.118.037655. PMID 30667281
- [Background] Dagan M, Dinh DT, Stehli J, Tan C, Brennan A, Warren J, Ajani AE, Freeman M, Murphy A, Reid CM, Hiew C, Oqueli E, Clark DJ, Duffy SJ. Sex disparity in secondary prevention pharmacotherapy and clinical outcomes following acute coronary syndrome. Eur Heart J Qual Care Clin Outcomes. 2022 Jun 6;8(4):420-428. doi: 10.1093/ehjqcco/qcab007. PMID 33537698
- [Background] Witt BJ, Jacobsen SJ, Weston SA, Killian JM, Meverden RA, Allison TG, Reeder GS, Roger VL. Cardiac rehabilitation after myocardial infarction in the community. J Am Coll Cardiol. 2004 Sep 1;44(5):988-96. doi: 10.1016/j.jacc.2004.05.062. PMID 15337208
- [Background] Crnko S, Du Pre BC, Sluijter JPG, Van Laake LW. Circadian rhythms and the molecular clock in cardiovascular biology and disease. Nat Rev Cardiol. 2019 Jul;16(7):437-447. doi: 10.1038/s41569-019-0167-4. PMID 30796369
- [Background] Heras M. [Ischemic heart disease in women: clinical presentation, non-invasive testing and management of acute coronary syndromes]. Rev Esp Cardiol. 2006 Apr;59(4):371-81. Spanish. PMID 16709390
- [Background] Hamood H, Hamood R, Green MS, Almog R. Determinants of adherence to evidence-based therapy after acute myocardial infarction. Eur J Prev Cardiol. 2016 Jun;23(9):975-85. doi: 10.1177/2047487315597209. Epub 2015 Jul 21. PMID 26198723
- [Background] Zhu B, Zhao Z, McCollam P, Anderson J, Bae JP, Fu H, Zettler M, Lenarz L. Factors associated with clopidogrel use, adherence, and persistence in patients with acute coronary syndromes undergoing percutaneous coronary intervention. Curr Med Res Opin. 2011 Mar;27(3):633-41. doi: 10.1185/03007995.2010.551657. Epub 2011 Jan 18. PMID 21241206
- [Background] Lewey J, Shrank WH, Bowry AD, Kilabuk E, Brennan TA, Choudhry NK. Gender and racial disparities in adherence to statin therapy: a meta-analysis. Am Heart J. 2013 May;165(5):665-78, 678.e1. doi: 10.1016/j.ahj.2013.02.011. Epub 2013 Mar 26. PMID 23622903
- [Background] Kumbhani DJ, Fonarow GC, Cannon CP, Hernandez AF, Peterson ED, Peacock WF, Laskey WK, Pan W, Schwamm LH, Bhatt DL; Get With the Guidelines Steering Committee and Investigators. Predictors of adherence to performance measures in patients with acute myocardial infarction. Am J Med. 2013 Jan;126(1):74.e1-9. doi: 10.1016/j.amjmed.2012.02.025. Epub 2012 Aug 24. PMID 22925314
- [Background] Bots SH, Inia JA, Peters SAE. Medication Adherence After Acute Coronary Syndrome in Women Compared With Men: A Systematic Review and Meta-Analysis. Front Glob Womens Health. 2021 Feb 22;2:637398. doi: 10.3389/fgwh.2021.637398. eCollection 2021. PMID 34816194
- [Background] Sakalaki M, Barywani S, Rosengren A, Bjorck L, Fu M. Determinants of suboptimal long-term secondary prevention of acute myocardial infarction: the structural interview method and physical examinations. BMC Cardiovasc Disord. 2019 Nov 6;19(1):243. doi: 10.1186/s12872-019-1238-5. PMID 31694556
- [Background] Marques-Vidal P, Jankowski P, De Bacquer D, Kotseva K; EUROASPIRE V collaborators. Dietary measures among patients with coronary heart disease in Europe. ESC EORP Euroaspire V. Int J Cardiol. 2020 Mar 1;302:5-14. doi: 10.1016/j.ijcard.2019.12.064. Epub 2019 Dec 31. PMID 31937454
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967
- [Background] Agewall S, Beltrame JF, Reynolds HR, Niessner A, Rosano G, Caforio AL, De Caterina R, Zimarino M, Roffi M, Kjeldsen K, Atar D, Kaski JC, Sechtem U, Tornvall P; WG on Cardiovascular Pharmacotherapy. ESC working group position paper on myocardial infarction with non-obstructive coronary arteries. Eur Heart J. 2017 Jan 14;38(3):143-153. doi: 10.1093/eurheartj/ehw149. No abstract available. PMID 28158518
- [Background] Schmidt S, Vilagut G, Garin O, Cunillera O, Tresserras R, Brugulat P, Mompart A, Medina A, Ferrer M, Alonso J. [Reference guidelines for the 12-Item Short-Form Health Survey version 2 based on the Catalan general population]. Med Clin (Barc). 2012 Dec 8;139(14):613-25. doi: 10.1016/j.medcli.2011.10.024. Epub 2012 Jan 11. Spanish. PMID 22244683
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Cantero MC, López-Roig S, Rodríguez-Marín J, Gelabert M, Pastor M-Á, Reig MT. Propiedades psicométricas de la Escala Hospitalaria de Ansiedad y Estrés (HAD) en población española. Ansiedad y Estrés. 2007;13:163-176
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Martin-Carrasco M, Otermin P, Perez-Camo V, Pujol J, Aguera L, Martin MJ, Gobartt AL, Pons S, Balana M. EDUCA study: Psychometric properties of the Spanish version of the Zarit Caregiver Burden Scale. Aging Ment Health. 2010 Aug;14(6):705-11. doi: 10.1080/13607860903586094. PMID 20544413
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC National Cardiac Societies; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur Heart J. 2021 Sep 7;42(34):3227-3337. doi: 10.1093/eurheartj/ehab484. No abstract available. PMID 34458905
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Schroder H, Fito M, Estruch R, Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Lamuela-Raventos R, Ros E, Salaverria I, Fiol M, Lapetra J, Vinyoles E, Gomez-Gracia E, Lahoz C, Serra-Majem L, Pinto X, Ruiz-Gutierrez V, Covas MI. A short screener is valid for assessing Mediterranean diet adherence among older Spanish men and women. J Nutr. 2011 Jun;141(6):1140-5. doi: 10.3945/jn.110.135566. Epub 2011 Apr 20. PMID 21508208
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Bueno H, Bernal JL, Jimenez-Jimenez V, Martin-Sanchez FJ, Rossello X, Moreno G, Goni C, Gil V, Llorens P, Naranjo N, Jacob J, Herrero-Puente P, Garrote S, Silla-Castro JC, Pocock SJ, Miro O; ICA-SEMES ad hoc COHERENT study group. The Clinical outcomes, healthcare resource utilization, and related costs (COHERENT) model. Application in heart failure patients. Rev Esp Cardiol (Engl Ed). 2022 Jul;75(7):585-594. doi: 10.1016/j.rec.2021.08.009. Epub 2021 Oct 20. English, Spanish. PMID 34688580
- [Result] Raparelli V, Norris CM, Bender U, Herrero MT, Kautzky-Willer A, Kublickiene K, El Emam K, Pilote L; GOING-FWD Collaborators. Identification and inclusion of gender factors in retrospective cohort studies: the GOING-FWD framework. BMJ Glob Health. 2021 Apr;6(4):e005413. doi: 10.1136/bmjgh-2021-005413. PMID 33836996

DOCUMENTS (1):
  • Study Protocol (2022-05-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT05619601/Prot_000.pdf